CLINICAL TRIAL: NCT05194007
Title: A Pilot Randomized, Double-blind, Placebo-controlled Trial to Investigate the Anti-inflammatory Effects of Frondanol in Adults With Inflammatory Bowel Disease
Brief Title: Investigating the Anti-inflammatory Effects of Frondanol in Adults With Inflammatory Bowel Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mohammed Bin Rashid University of Medicine and Health Sciences (Other)
Collaborators: Mediclinic Middle East (Industry); Rashid Hospital (Other Government); Dubai Health Authority (Other Government)
Responsible Party: Principal Investigator, Reem Jan, Assistant Professor, Mohammed Bin Rashid University of Medicine and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2021-11-18; First posted 2022-01-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Ulcerative Colitis Chronic Mild; Ulcerative Colitis Chronic Moderate; Crohn Colitis
Keywords: inflammatory bowel disease; Crohn disease; ulcerative colitis; frondanol; randomized controlled trial; placebo-controlled; chronic bowel inflammation
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Colitis, Ulcerative | interventions — Frondanol-A5P

STUDY DESIGN:
Intervention Model Description: This is a parallel group, randomized, double-blind, placebo-controlled pilot trial where participants will be randomized to receive either Frondanol 1000mg twice daily or placebo twice daily for 6 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All patients and investigators, excluding the study coordinator, will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental -Frondanol (Experimental): Eligible participants will receive Frondanol capsule orally (1000 mg capsule twice daily) for 6 months
  Interventions: Drug: Frondanol
- Placebo (Placebo Comparator): Eligible participants will receive placebo capsule (twice daily) for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Frondanol — Frondanol capsule (1000 mg) will be administered orally (Twice daily) in the double blind settings
  Arms: Experimental -Frondanol
Drug: Placebo — Placebo (corn starch) capsule will be administered orally (Twice daily) in the double blind settings
  Arms: Placebo

SUMMARY:
This is a pilot, prospective, double-blinded, two-arm, randomized controlled trial of the efficacy of Frondanol in comparison to placebo in decreasing bowel inflammation in patients with a clinical diagnosis of inflammatory bowel disease who are in remission and on standard of care treatment.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD), consisting of Crohn's disease and ulcerative colitis, is a debilitating condition, particularly during active periods (flares) of the disease and can sometimes lead to life-threatening complications. IBD is characterized by chronic gut inflammation resulting in symptoms such as severe diarrhea, abdominal pain, blood in stool, fatigue and unintended weight loss, which significantly affect the quality of life of patients. Although the exact mechanism underlying the chronic gut inflammation is not fully understood, several cytokine networks are thought to be involved. Currently, treatment of IBD relies on minimizing symptoms and improving quality of life through the control of disease progression and complications; however, these drugs have significant systemic side effects that reduce their tolerability. Moreover, up to 40% of patients still exhibit non-response to therapy, and these treatment-refractory patients would require alternative therapeutic approaches. Frondanol, a widely available nutraceutical extract of the edible sea cucumber, Cucumaria frondosa, has been reported to possess potent anti-inflammatory effects in both animals and humans, whilst showing no signs of toxicity. The potent anti-inflammatory effects of Frondanol in a mouse model of IBD provide encouragement for investigating its effects in human IBD patients. The proposed study is a pilot, double-blinded, placebo-controlled trial of Frondanol in patients with IBD (Crohn's disease or ulcerative colitis) who are currently in remission and are on standard therapy. One hundred patients will be randomized (1:1) to receive Frondanol or placebo as an adjunct to their standard therapy for the period of six months. Blood and tissue samples from colon biopsies obtained during routine visits and endoscopies at baseline and six months later will be collected. The levels of inflammatory markers such as myeloperoxidase, tumor necrosis factor (TNF)-α, interleukin (IL)1β, IL6, IL17A, IL22, interferon gamma (IFN-γ) and several other inflammatory markers will be compared between patients treated with Frondanol and those treated with placebo, and the findings will be correlated with clinical and histological parameters. Over the past 25 years, it is estimated that more than 3 million Frondanol capsules have been consumed on the human market with no reported side effects. An even larger amount has been consumed on the veterinary market without a single reported incident. If proven beneficial, Frondanol, will be a useful supplement in treating the underlying chronic gut inflammation in IBD patients, increasing the likelihood of patients remaining in remission and potentially providing an effective, natural and safe treatment for treatment naive patients in the future.

ELIGIBILITY:
Inclusion criteria:

* A confirmed clinical diagnosis of IBD of any duration, age 18 years or older, with mild to moderate disease and on standard therapy.
* The diagnostic criteria for IBD include the presence of chronic diarrhea for more than four weeks, and evidence of active inflammation on endoscopy and chronic changes on biopsy.
* Patients with stable mild to moderate IBD will be eligible for the study.
* Stable IBD is defined as having stable symptoms over a period of several weeks, diagnostic evaluation has been completed and the patient has been on consistent medication.
* Mild to moderate IBD is indicated by a Partial Mayo score (Mayo Clinic Score/Disease Activity Index for Colitis) of between 1-6, and a total of Mayo score of 1-10.
* For patients with Crohn's disease, only those with Crohn's colitis will be included (patients with small bowel disease are eligible to enter the trial as long as they also have large bowel inflammation).

Exclusion criteria:

* Pregnancy, breastfeeding, allergy to seafood or marine products
* Severe medical illness such as uncontrolled diabetes (HbA1C>10), significant or unstable cardiovascular or pulmonary disease, impaired renal function (Cr>2.0mg/dL), current or recent (<1 year) malignancy, or other significant medical illness that in the view of the investigators may impair participation in the study.
* Patients with severe IBD (defined by a Partial Mayo score of 7-9 and a total Mayo score of 11-12, with active symptoms) will not be eligible to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-02-19 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
To assess the change in plasma levels of cytokines between IBD patients treated with Frondanol and those treated with placebo at baseline and after six months of treatment | Baseline and after 6 months
  Cytokines will be measured in plasma samples.
To assess the change in plasma levels of marker of inflammation between IBD patients treated with Frondanol and those treated with placebo at baseline and after six months of treatment | Baseline and after 6 months
  Marker of inflammation will be measured in plasma samples.
To assess the change in biopsy mRNA levels between IBD patients treated with Frondanol and those treated with placebo at baseline and after six months of treatment | Baseline and after 6 months
  The mRNA levels of transcription factors involved in inflammation will be measured in tissue biopsy samples
To assess the change in the biopsy mRNA levels between IBD patients treated with Frondanol and those treated with placebo at baseline and after six months of treatment | Baseline and after 6 months
  The mRNA levels of cytokines involved in inflammation will be measured in tissue biopsy samples
To assess the change in the biopsy mRNA levels between IBD patients treated with Frondanol and those treated with placebo at baseline and after six months of treatment | Baseline and after 6 months
  The mRNA levels of markers involved in inflammation will be measured in tissue biopsy samples
To assess the change in the proteins expression between IBD patients treated with Frondanol and those treated with placebo at baseline and after six months of treatment | Baseline and after 6 months
  The proteins expression of transcription factors involved in inflammation will be measured in tissue biopsy samples
To assess the change in the proteins expression between IBD patients treated with Frondanol and those treated with placebo at baseline and after six months of treatment | Baseline and after 6 months
  The proteins expression cytokines involved in inflammation will be measured in tissue biopsy samples
To assess the change in the proteins expression between IBD patients treated with Frondanol and those treated with placebo at baseline and after six months of treatment | Baseline and after 6 months
  The proteins expression of markers involved in inflammation will be measured in tissue biopsy samples

SECONDARY OUTCOMES:
To assess the change in routine clinical parameters between IBD patients treated with Frondanol and those treated with placebo at baseline and after six months of treatment: | Baseline and after 2 months and after 4 months and after 6 months
  Mayo score, which are based on ratings of frequency and severity of clinical symptoms and endoscopic activity will be measured.
To assess the change in routine clinical parameters between IBD patients treated with Frondanol and those treated with placebo at baseline and after six months of treatment: | Baseline and after 2 months and after 4 months and after 6 months
  Complete blood count will be measured
To assess the change in routine clinical parameters between IBD patients treated with Frondanol and those treated with placebo at baseline and after six months of treatment: | Baseline and after 2 months and after 4 months and after 6 months
  Erythrocyte sedimentation rate will be measured
To assess the change in routine clinical parameters between IBD patients treated with Frondanol and those treated with placebo at baseline and after six months of treatment: | Baseline and after 2 months and after 4 months and after 6 months
  Serum C-reactive protein will be measured
To assess the change in routine clinical parameters between IBD patients treated with Frondanol and those treated with placebo at baseline and after six months of treatment: | Baseline and after 2 months and after 4 months and after 6 months
  Serum albumin will be measured
To assess the change in routine clinical parameters between IBD patients treated with Frondanol and those treated with placebo at baseline and after six months of treatment: | Baseline and after 2 months and after 4 months and after 6 months
  Fecal calprotectin will be measured

CONTACTS AND LOCATIONS:
Locations (2):
- United Arab Emirates (2):
  - Mediclinic City Hospital, Dubai
  - Mediclinic Parkview Hospital, Dubai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaser A, Zeissig S, Blumberg RS. Inflammatory bowel disease. Annu Rev Immunol. 2010;28:573-621. doi: 10.1146/annurev-immunol-030409-101225. PMID 20192811
- [Background] Molodecky NA, Soon IS, Rabi DM, Ghali WA, Ferris M, Chernoff G, Benchimol EI, Panaccione R, Ghosh S, Barkema HW, Kaplan GG. Increasing incidence and prevalence of the inflammatory bowel diseases with time, based on systematic review. Gastroenterology. 2012 Jan;142(1):46-54.e42; quiz e30. doi: 10.1053/j.gastro.2011.10.001. Epub 2011 Oct 14. PMID 22001864
- [Background] Ng SC, Shi HY, Hamidi N, Underwood FE, Tang W, Benchimol EI, Panaccione R, Ghosh S, Wu JCY, Chan FKL, Sung JJY, Kaplan GG. Worldwide incidence and prevalence of inflammatory bowel disease in the 21st century: a systematic review of population-based studies. Lancet. 2017 Dec 23;390(10114):2769-2778. doi: 10.1016/S0140-6736(17)32448-0. Epub 2017 Oct 16. PMID 29050646
- [Background] Friedrich M, Pohin M, Powrie F. Cytokine Networks in the Pathophysiology of Inflammatory Bowel Disease. Immunity. 2019 Apr 16;50(4):992-1006. doi: 10.1016/j.immuni.2019.03.017. PMID 30995511
- [Background] Kuhn KA, Schulz HM, Regner EH, Severs EL, Hendrickson JD, Mehta G, Whitney AK, Ir D, Ohri N, Robertson CE, Frank DN, Campbell EL, Colgan SP. Bacteroidales recruit IL-6-producing intraepithelial lymphocytes in the colon to promote barrier integrity. Mucosal Immunol. 2018 Mar;11(2):357-368. doi: 10.1038/mi.2017.55. Epub 2017 Aug 16. PMID 28812548
- [Background] Lee JS, Tato CM, Joyce-Shaikh B, Gulen MF, Cayatte C, Chen Y, Blumenschein WM, Judo M, Ayanoglu G, McClanahan TK, Li X, Cua DJ. Interleukin-23-Independent IL-17 Production Regulates Intestinal Epithelial Permeability. Immunity. 2015 Oct 20;43(4):727-38. doi: 10.1016/j.immuni.2015.09.003. Epub 2015 Sep 29. PMID 26431948
- [Background] Sairenji T, Collins KL, Evans DV. An Update on Inflammatory Bowel Disease. Prim Care. 2017 Dec;44(4):673-692. doi: 10.1016/j.pop.2017.07.010. Epub 2017 Oct 5. PMID 29132528
- [Background] Ben-Horin S, Chowers Y. Tailoring anti-TNF therapy in IBD: drug levels and disease activity. Nat Rev Gastroenterol Hepatol. 2014 Apr;11(4):243-55. doi: 10.1038/nrgastro.2013.253. Epub 2014 Jan 7. PMID 24393836
- [Background] Guerra I, Bermejo F. Management of inflammatory bowel disease in poor responders to infliximab. Clin Exp Gastroenterol. 2014 Sep 18;7:359-67. doi: 10.2147/CEG.S45297. eCollection 2014. PMID 25258548
- [Background] Kelly MS. Echinoderms: their culture and bioactive compounds. Prog Mol Subcell Biol. 2005;39:139-65. PMID 17152697
- [Background] Janakiram NB, Mohammed A, Bryant T, Lightfoot S, Collin PD, Steele VE, Rao CV. Improved innate immune responses by Frondanol A5, a sea cucumber extract, prevent intestinal tumorigenesis. Cancer Prev Res (Phila). 2015 Apr;8(4):327-37. doi: 10.1158/1940-6207.CAPR-14-0380. Epub 2015 Feb 5. PMID 25657017
- [Background] Janakiram NB, Mohammed A, Zhang Y, Choi CI, Woodward C, Collin P, Steele VE, Rao CV. Chemopreventive effects of Frondanol A5, a Cucumaria frondosa extract, against rat colon carcinogenesis and inhibition of human colon cancer cell growth. Cancer Prev Res (Phila). 2010 Jan;3(1):82-91. doi: 10.1158/1940-6207.CAPR-09-0112. PMID 20051375
- [Background] Subramanya SB, Chandran S, Almarzooqi S, Raj V, Al Zahmi AS, Al Katheeri RA, Al Zadjali SA, Collin PD, Adrian TE. Frondanol, a Nutraceutical Extract from Cucumaria frondosa, Attenuates Colonic Inflammation in a DSS-Induced Colitis Model in Mice. Mar Drugs. 2018 Apr 30;16(5):148. doi: 10.3390/md16050148. PMID 29710854
- [Derived] Ghelani H, Adrian TE, Ho SB, Akhras J, Azar AJ, Jan RK. Study protocol for a pilot randomized, double-blind, placebo-controlled trial to investigate the anti-inflammatory effects of Frondanol in adults with inflammatory bowel disease. Contemp Clin Trials Commun. 2022 Dec 1;31:101046. doi: 10.1016/j.conctc.2022.101046. eCollection 2023 Feb. PMID 36544548

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-04): https://cdn.clinicaltrials.gov/large-docs/07/NCT05194007/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-04): https://cdn.clinicaltrials.gov/large-docs/07/NCT05194007/ICF_001.pdf